CLINICAL TRIAL: NCT00889174
Title: Leukodystrophies of Unknown Cause
Brief Title: The Nosology and Etiology of Leukodystrophies of Unknown Causes
Status: Completed | Type: Observational
Sponsor: National Human Genome Research Institute (NHGRI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 090128; 09-HG-0128
Record Dates: First submitted 2009-04-25; First posted 2009-04-28 (Estimated); Last update posted 2018-08-03 (Actual); Status verified 2018-08-01

CONDITIONS: Leukodystrophy; Leukoencephalopathy
Keywords: Genetic Disorders of the White Matter; Leukodystrophies; Myelin; White Matter Disorder; Genetic Disorder
MeSH Terms: conditions — Leukoencephalopathies; Genetic Diseases, Inborn

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other

SUMMARY:
Background:

- A leukodystrophy is a disease affecting the white matter of the brain. The white matter conducts electricity from one part of the brain to the other. If the insulation, or myelin, is damaged, the brain s electrical pathways will not work properly. Researchers are trying to identify what causes leukodystrophy.

Objectives:

* To collect detailed clinical characterizations, including histories, physical examinations, biochemical tests, genetic studies, and neurophysiologic and neuroimaging studies in patients with unclassified leukodystrophies to comprehensively characterize such patients and obtain comparative clinical profiles.
* To collect detailed clinical characterizations, including histories, physical examinations, biochemical tests, genomic and proteomic tissue, and neurophysiologic and neuroimaging studies in patients with known leukodystrophies to investigate the underlying pathogenesis of these disorders.
* To better understand leukodystrophies of unknown cause and to identify the part of the DNA of the patient with leukodystrophy that is causing the problem.

Eligibility:

* Any individual with a known or suspected leukodystrophy is eligible to participate in this protocol, including

  * Patients with white matter disease that is unclassified or of unknown cause, including but not limited to leukoencephalopathies with calcifications, leukoencephalopathies with cysts, leukoencephalopathies with hypomyelination, and leukoencephalopathies with brainstem involvement.
  * Parents or siblings of these subjects.
* Exclusion criteria include patients too ill to travel to the Clinical Center and patients for whom the leukoencephalopathy is felt to be secondary to an acquired cause (for example, traumatic or infectious).

Design:

* Patients will be seen either as an inpatient or outpatient depending on the tests that are planned. Patients may need to stay at the Clinical Center for 3 to 5 days.
* The following tests will be conducted as part of standard clinical care:

  * Physical and neurological examinations, including blood and urine tests.
  * Magnetic resonance based studies to produce a picture of the patient s brain (under general anesthesia).
  * Spinal tap to measure chemicals in the spinal fluid (under general anesthesia in young children).
  * Nerve biopsy, if the peripheral nerves are affected, or muscle biopsy, if the cells called the mitochondria or the muscles are involved (both under general anesthesia).
* The following studies may be performed as part of participation in the research:

  * Blood, urine, spinal fluid, or muscle to understand the proteins, DNA, and molecules in these tissues.
  * Skin biopsy to grow (in culture) skin cells and to analyze the skin microscopically.
  * DNA studies to find new genes responsible for leukodystrophies and to better understand these diseases.
* Participation should be based on an interest to help further the research on leukodystrophies. Specific information about a patient s present or future health risks may not be gained.

DETAILED DESCRIPTION:
Genetic white matter disorders (leukodystrophies) are estimated to have an incidence of 1:5000 live births. As many as 50% of patients with white matter disease remain undiagnosed after conventional neuroimaging, biochemical and genetic testing, and therefore have unclassified leukodystrophies. Moreover, the mechanisms of disease in many leukodystrophies of known cause are very poorly understood: many are systemic abnormalities that manifest only in white matter. The purpose of this study is to: (a) define novel homogeneous groups of patients with leukodystrophy and work toward finding the cause of these disorders and (b) establish disease mechanisms in selected classified leukodystrophies. In order to achieve these goals, patients with leukodystrophy will be analyzed by clinical, neurophysiological, biochemical and genetic means. For goal (a), patients would have been diagnosed as having an unclassified leukodystrophy or no known cause of their leukodystrophy at outside centers. At the Clinical Center, such patients will undergo a series of neuropsychological, blood, urine, spinal fluid, radiological, and peripheral tissue pathological tests. Some of these tests will be part of a standard battery while others will be tailored to individual patients. For goal (b), selected leukodystrophies with a defined genetic cause will be selected for further mechanistic study, using clinical and laboratory tools to establish increased understanding of the underlying pathophysiology. It is hoped that the present study will help clarify the nosology of the leukodystrophies and significantly advance our understanding of the pathogenesis of these diseases.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Patients with white matter disease that is unclassified or of unknown cause, including, but not limited to leukoencephalopathies with calcifications, leukoencephalopathies with cysts, leukoencephalopathies with hypomyelination and leukoencephalopathies with brainstem involvement.
* Parents or siblings of these subjects

EXCLUSION CRITERIA:

* Patients meeting above criteria but too ill to travel to the clinical center. In that case, consideration will be given to enrolling them for the collection of medical records and samples only.
* Patients meeting above criteria, but where the leukoencephalopathy is felt to be secondary to an acquired cause, for example traumatic or infectious.

Ages: 1 Month to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2009-04-24; Study Completion 2018-08-01

CONTACTS AND LOCATIONS:
Overall Officials: William A Gahl, M.D., Principal Investigator — National Human Genome Research Institute (NHGRI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Linnankivi TT, Autti TH, Pihko SH, Somer MS, Tienari PJ, Wirtavuori KO, Valanne LK. 18q-syndrome: brain MRI shows poor differentiation of gray and white matter on T2-weighted images. J Magn Reson Imaging. 2003 Oct;18(4):414-9. doi: 10.1002/jmri.10383. PMID 14508777
- [Background] Gay CT, Hardies LJ, Rauch RA, Lancaster JL, Plaetke R, DuPont BR, Cody JD, Cornell JE, Herndon RC, Ghidoni PD, Schiff JM, Kaye CI, Leach RJ, Fox PT. Magnetic resonance imaging demonstrates incomplete myelination in 18q- syndrome: evidence for myelin basic protein haploinsufficiency. Am J Med Genet. 1997 Jul 25;74(4):422-31. doi: 10.1002/(sici)1096-8628(19970725)74:43.0.co;2-k. PMID 9259379
- [Background] Ugur SA, Tolun A. A deletion in DRCTNNB1A associated with hypomyelination and juvenile onset cataract. Eur J Hum Genet. 2008 Feb;16(2):261-4. doi: 10.1038/sj.ejhg.5201935. Epub 2007 Oct 10. PMID 17928815